CLINICAL TRIAL: NCT03517761
Title: A Single-Blinded, Randomized Controlled Trial Evaluating the Use of Bone Marrow Concentrate for the Treatment of Alar, Accessory, and Transverse Ligament Injuries
Brief Title: Use of Bone Marrow Concentrate for Treatment of Alar, Accessory, and Transverse Ligament Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RSI2017-RCT01
Record Dates: First submitted 2018-03-23; First posted 2018-05-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Craniocervical Injuries
Keywords: CCJ; Bone Marrow Concentrate; Stem Cell Therapy; Alar Ligament; Transverse Ligament
MeSH Terms: conditions — Trauma, Nervous System

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, single-blinded, randomized, controlled study to include 80 subjects total, 40 treated with Bone Marrow Concentrate and 40 subjects treated with a Sham Procedure with cross-over from the sham to active group at 6 months
Who Masked: Participant
Masking Description: Participants are blind to treatment condition until 6 months post-procedure. Participants in sham control group can crossover to treatment group at that time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bone Marrow Concentrate treatment (Experimental): Bone marrow concentrate subjects will undergo a bone marrow aspiration of approximately 30-60 cc. Platelet rich plasma (PRP) and platelet lysate (PL) will be derived from the bone marrow aspirate and later mixed with the bone marrow nucleated cell layer. Injectate will then be used to treat the ligaments in the CCJ and upper cervical injections to C0-C3 ligaments and facets.
  Interventions: Biological: Bone Marrow Concentrate treatment
- Sham Control (Sham Comparator): Control subjects will also undergo a bone marrow aspiration of 30-60 cc to maintain blinding. Control subjects will receive a sham procedure of a small skin puncture to the posterior oropharynx guided under fluoroscopy while under anesthesia as well as receive sham upper cervical injections to C0-C3 ligaments and facets.
  Interventions: Other: Sham Control

INTERVENTIONS:
Biological: Bone Marrow Concentrate treatment — While under unconscious TIVA anesthesia, the injectate is then injected under fluoroscopy into the area in need of treatment using an anterior approach through the posterior oropharynx with direct visualization of the injection site via endoscopy. The alar, transverse, and accessory ligaments are the target areas to be treated with the bone marrow concentrate injectate. Patients will be repositioned in the prone position to then receive upper cervical injections to C0-C3 ligaments and facets.Patients will receive 2 of these treatment procedures 3 months apart.
  Arms: Bone Marrow Concentrate treatment
Other: Sham Control — Control subjects will receive a sham procedure of a small skin puncture to the posterior oropharynx guided under fluoroscopy while under anesthesia.Patients will also receive small skin punctures to the back of the neck to mimic ligament and facet injections. Patients will receive 2 of these procedure 3 months apart.
  Arms: Sham Control

SUMMARY:
The purpose of this study is to evaluate the effectiveness of using anterior approach through the posterior oropharynx for treating alar and transverse ligament injuries with bone marrow concentrate for patients with craniocervical junction (CCJ) instability.

DETAILED DESCRIPTION:
This study will be a single-center, prospective, single-blinded, randomized, controlled study of patients with CCJ instability that are randomized to either 2 bone marrow concentrate (BMC) treatments or 2 sham procedure to evaluate the safety and effectiveness of using an anterior approach through the posterior oropharynx for treating alar and transverse ligament injuries in addition to upper cervical injection treatment. Patients will undergo a bone marrow aspiration of approximately 30-60 cc from the posterior superior iliac crest for each procedure. Platelet rich plasma (PRP) and platelet lysate (PL) will be derived from the bone marrow aspirate and later mixed with the bone marrow nucleated cell layer for those in the treatment group. While under unconscious TIVA anesthesia, the injectate is then injected under fluoroscopy into the area in need of treatment using an anterior approach through the posterior oropharynx with direct visualization of the injection site via endoscopy. Patients will be repositioned in the prone position to then receive upper cervical injections to C0-C3 ligaments and facets. Patients assigned to the sham control condition will also undergo a bone marrow aspiration of 30-60 cc to maintain blinding. Control subjects will receive a sham procedure of a small skin puncture to the posterior oropharynx guided under fluoroscopy while under anesthesia, as well as those pokes to mimic the upper cervical injections to the C0-C3 ligaments and facets. In this group, the BMC will be donated for research purposes and not used clinically. Study patients will be evaluated at 3 months after the 2nd procedure months using patient reported clinical outcome questionnaires and digital motion x-ray. Control patients can crossover to the treatment group after being unblinded at 3-months after the 2nd procedure.

As an alternative to invasive surgery, ligament injections of proliferant agents (prolotherapy) have been proposed to treat cervical instability. Our group has used a blinded flexion-extension radiography to demonstrate that injections of cervical proliferant agents (hypertonic dextrose) into the supraspinous and interspinous ligaments can objectively reduce excessive cervical translation in flexion (Centeno et al. 2005). More recently we have published on the use of bone marrow concentrate to demonstrate MRI evidence of robust ACL ligament signal changes consistent with healing and repair (Centeno et al. 2015).

One of the challenges of treating the upper cervical ligaments through injection is that they can't be accessed from the posterior due to obstruction from the cervical spinal cord.Our group has developed an injection technique using an anterior approach through the posterior oropharynx, which allows direct access to the ligaments for injection. The goal of this study is to evaluate the effectiveness of this procedure in carefully selected CCJ instability patients.

ELIGIBILITY:
Inclusion Criteria:

-1) Voluntary signature of the IRB approved Informed Consent, 2) Skeletally mature Male or Female ages 18 to 65 3) Must have a specific inciting injury event that occurred less than 10 years ago where the patient experienced trauma that caused the problem-meaning from that day on, they had the symptoms for which they are now seeking treatment 4) Upper cervical symptoms predominate: Patient must have a headache since the event and must have one of the following: dizziness, vertigo, imbalance, or visual disturbances 5) Patient must be able to care for themselves without assistance 6) NDI percentage score (raw NDI score times 2) at least 30 (moderate disability) 7) Imaging: Must have DMX lateral overhang of C1 on C2 in lateral bending open mouth view of at least 3mm or grabb-oakes of >9mm on cervical flexion MRI-change in signal on static imaging does not qualify the patient 8) Has not responded long-term to conservative care 9) Upper cervical fusion candidate 10) Exam is c/w upper cervical injury (i.e. tenderness along upper cervical facet joints and/or musculature/skull base, proprioceptive difficulties)

11) Is independent, ambulatory, and can comply with all post-operative evaluations and visits 12) Patient states strong desire to avoid surgery

Exclusion criteria:

13) Known or diagnosed EDS based on Beighton criteria: https://www.physio-pedia.com/Beighton_score 14) Lower or mid-cervical symptomatic disease (tenderness in mid to lower cervical facets, radiculopathy, radiating symptoms into shoulder blade, epicondylitis, numbness and tingling in hands) 15) Prior spinal fusion or surgery at any segment in cervical, thoracic, or lumbar spine 16) NDI % score > than 56 (severe disability), unless at the discretion of the independent physician review 17) Prior or current history of a metabolic disorder like diabetes, anorexia, other eating disorder, BMI>40 18) Unable to tolerate injections due to central sensitization (i.e. significant intolerance to manual therapy such as massage, activity such as physical therapy, or an exaggerated pain response to prior injection therapy) 19) Prior epidural or other milligram dose steroid injection in any area within the past 6 months 20) Prior prolotherapy or platelet-based injections to the cervical spine within the last 3 months 21) Prior radiofrequency ablation to the cervical spine within the last 2 years 22) Physical infirmity that is incompatible with the procedure and/or anesthesia required for same 23) Unable to tolerate the injection position 24) Abnormal anatomy seen on MRI imaging that would make the procedure higher risk (e.g. congenital atlanto-axial fusion, atlas assimilation, upper cervical fracture or surgical fusion) 25) Inflammatory or auto-immune based pathology (e.g., rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis, polymyalgia, polymyositis, gout, pseudo gout) 26) Quinolone or Statin induced myopathy/tendinopathy 27) Condition represents a worker's compensation case 28) Currently involved in a health-related litigation procedure 29) Is pregnant 30) Bleeding disorders 31) Currently taking anticoagulant or immunosuppressive medication 32) Allergy or intolerance to study medication 33) Use of and significant physical dependence on a chronic opioid (>20 mg oxycodone equivalent per day) 34) Documented history of drug abuse within six months of treatment 35) Any other condition, that in the opinion of the investigator, that would preclude the patient from enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-03-23 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Headache Impact Test score change from baseline | Change from Baseline to 3 months after 2nd treatment
  The difference between treatment groups in the within patient mean change from baseline to 6 months in Headache Impact Test scores.

SECONDARY OUTCOMES:
Neck Disability Index score change from baseline | Change from baseline to 3 months after 2nd treatment
  Difference between groups in changes scores for Neck Disability Index scores from baseline and 6 months.
Neck Disability Index score change from baseline | Change from baseline to 6 months after 2nd treatment
  Difference between groups in changes scores for Neck Disability Index scores from baseline and 12 months.
Short Form Health Survey change from baseline | Change from baseline to 3 months after 2nd treatment
  Difference between groups in changes scores for Short Form Health Survey scores from baseline and 6 months.
Short Form Health Survey change from baseline | Change from baseline to 6 months after 2nd treatment
  Difference between groups in changes scores for Short Form Health Survey scores from baseline and 12 months.
Numeric Pain Scale change from baseline | Change from baseline to 3 months after 2nd treatment
  Difference between groups in changes scores for numeric pain scores from baseline and 6 months, where 0=no pain and 10=worst possible pain.
Numeric Pain Scale change from baseline | Change from baseline to 6 months after 2nd treatment
  Difference between groups in changes scores for numeric pain scores from baseline and 12 months, where 0=no pain and 10=worst possible pain.
Single Assessment Numeric Evaluation improvement rating -modified | mean at 3 months after 2nd treatment
  Difference between groups for mean improvement scores at 6 months, where -100=100% worse from baseline and 100=100% better or improved from baseline
Single Assessment Numeric Evaluation improvement rating -modified | mean at 6 months after 2nd treatment
  Difference between groups for mean improvement scores at 12 months, where -100=100% worse from baseline and 100=100% better or improved from baseline
Adverse events | Thru 6 month post procedure after 2nd treatment
  Any complication of adverse event
C1-C2 overhang | 3 months after 2nd treatment
  Post-op DMX studies will also be used to quantify any reduction in C1-C2 overhang or ADI.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Centeno, MD, Principal Investigator — Regenexx, LLC
Locations (1):
- Ehren Dodson, Broomfield, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centeno CJ, Elliott J, Elkins WL, Freeman M. Fluoroscopically guided cervical prolotherapy for instability with blinded pre and post radiographic reading. Pain Physician. 2005 Jan;8(1):67-72. PMID 16850045
- [Background] Panjabi MM, Crisco JJ 3rd, Lydon C, Dvorak J. The mechanical properties of human alar and transverse ligaments at slow and fast extension rates. Clin Biomech (Bristol). 1998 Mar;13(2):112-120. doi: 10.1016/s0268-0033(97)00053-3. PMID 11415778
- [Background] Rajwanshi A, Rohilla M, Singh P. Trans-oral fine needle aspiration cytology in cervical (C1 and C2) vertebral lesions: a novel diagnostic approach. Cytopathology. 2017 Feb;28(1):31-34. doi: 10.1111/cyt.12361. Epub 2016 Aug 3. PMID 27489015
- [Background] Centeno CJ, Pitts J, Al-Sayegh H, Freeman MD. Anterior cruciate ligament tears treated with percutaneous injection of autologous bone marrow nucleated cells: a case series. J Pain Res. 2015 Jul 31;8:437-47. doi: 10.2147/JPR.S86244. eCollection 2015. PMID 26261424